CLINICAL TRIAL: NCT00714324
Title: Validation of Nutritional Screening for Patient Use
Brief Title: Simplified Nutritional Screening for Patient Use
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Southampton (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Christine McGrath, Southampton University Hospitals NHS trust
Other Study IDs: ELIA003
Record Dates: First submitted 2008-07-03; First posted 2008-07-14 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Malnutrition
Keywords: Nutrition; Screening
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Paper screening
- 2: Electronic screening

SUMMARY:
The purpose of this study is to determine if patients are able to reliably screen themselves for nutrition risk.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Adults aged > 18years
* Able to complete screening and provide written informed consent
* Willingness to take part

Exclusion Criteria:

* Children (<18years)
* Pregnant women
* Inpatients
* Unable to complete screen due to physical or mental incapacity
* Unable to comprehend oral and written English language
* Participation in other nutrition studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending general outpatient clinics
Sampling Method: Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
To validate the use of a screening tool for patient use | 1 year

SECONDARY OUTCOMES:
To assess prevalence of malnutrition in outpatients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marinos Elia, Professor, Principal Investigator — University of Southampton
Locations (1):
- Southampton University Hospitals NHS trust, Southampton, Hampshire, United Kingdom

REFERENCES:
- [Derived] Cawood AL, Elia M, Sharp SK, Stratton RJ. Malnutrition self-screening by using MUST in hospital outpatients: validity, reliability, and ease of use. Am J Clin Nutr. 2012 Nov;96(5):1000-7. doi: 10.3945/ajcn.112.037853. Epub 2012 Oct 3. PMID 23034963